CLINICAL TRIAL: NCT01288781
Title: Intracranial Pressure in Experimental Models of Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangor University (Other)
Collaborators: Universita di Verona (Other); North Wales Research Committee, UK (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: F002686; 2010-019520-31 (EudraCT Number)
Record Dates: First submitted 2011-01-27; First posted 2011-02-02 (Estimated); Results first posted 2011-12-26 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2011-12

CONDITIONS: High Altitude Headache
Keywords: High Altitude Headache; intra-cranial pressure; hypoxia
MeSH Terms: conditions — Hypoxia | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetazolamide (Experimental): Arm 1: ACETAZOLAMIDE (250mg) will be given to subjects at fifteen, twenty and thirty two hours post hypoxic exposure (3777m).
  Interventions: Drug: Acetazolamide
- Placebo (Placebo Comparator): Placebo (LACTOSE MONOHYDRATE) will be given to subjects at fifteen, twenty and thirty two hours post hypoxic exposure (3777m).
  Interventions: Drug: Lactose monohydrate

INTERVENTIONS:
Drug: Acetazolamide — During a forty eight hour hypoxic exposure (3777m), subjects will be given either acetazolamide or placebo at hours fifteen, twenty and thirty two.
  Other Names: Diamox
  Arms: Acetazolamide
Drug: Lactose monohydrate — During a forty eight hour hypoxic exposure (3777m), subjects will be given either acetazolamide or placebo at hours fifteen, twenty and thirty two.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether increased pressure in the head is elevated in people who suffer from High Altitude Headache. We hypothesise that head pressure will be elevated in people with High Altitude Headache.

DETAILED DESCRIPTION:
High Altitude Headache is the primary symptom of Acute Mountain Sickness. However, at present the reason why some individuals suffer from High Altitude Headache and others do not remains unknown. It is widely believed that elevated pressure within the brain leads to stretching of pain sensitive fibres and thus headache. However, evidence of raised intracranial pressure during High Altitude Headache is currently unavailable. Therefore, this study aims to examine a proxy measure of intracranial pressure (Optic Nerve Sheath Diameter) in persons visiting High Altitude, half of whom have been given the drug acetazolamide that is known to reduce headache symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Member of the Italian High Altitude Research Expeditions

Exclusion Criteria:

* Are under the age of 18years;
* sulfonamide allergy
* Liver or kidney disfunction
* Have any other uncontrolled medical condition
* Or are unable to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin S Lawley, BSc, Principal Investigator — Bangor University
Locations (1):
- School of Sport, Health and Exercise Sciences, Bangor University, Bangor, Gwynedd, United Kingdom

REFERENCES:
- [Derived] Lawley JS, Oliver SJ, Mullins P, Morris D, Junglee NA, Jelleyman C, Macdonald JH. Optic nerve sheath diameter is not related to high altitude headache: a randomized controlled trial. High Alt Med Biol. 2012 Sep;13(3):193-9. doi: 10.1089/ham.2012.1019. PMID 22994519

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants attending the Antur Ymchwil 2011 Expedition to the European Alps were recruited between 01.07.11 and 01.08.11.
Pre-assignment Details: Participants completed two trials, including a 12 hour sea level exposure followed by a 36 hour high altitude exposure (3777m). Participants were assigned to one of two groups based on High-altitude headache susceptibility determined by visual analogue score obtained after 12 hours at high altitude. No participants were excluded.
Period: Overall Study
Arm/Group | Acetazolamide | Placebo
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetazolamide | Placebo | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24 (6) | 20 (1) | 21 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United Kingdom | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Optic Nerve Sheath Diameter by Ultrasonography
Description: Baseline is defined as the average of the 3 hour and 12 hour normoxia measurement.
  24 hours is defined at the 24 hour hypoxia measurement. Optic nerve sheath diameter obtained by ultrasonography of the eye. Increased optic nerve sheath diameter suggests greater intra cranial pressure.
Time Frame: Optic Nerve Sheath Diameter: baseline, 24 hours.
Population: All participants were included. Analysis was intention to treat. There were no missing data.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 11 | 12
mm | 0.02 (0.06) | 0.02 (0.06)
Statistical Analysis 1: Comparison: Acetazolamide vs Placebo; Omnibus analysis was performed. 2 (drug: Acetazolamide versus placebo) * 2 (susceptibility: high altitude headache resistant versus high altitude headache susceptible) * 6 (time: sea level, 3 & 12; high altitude, 3, 12, 24 & 36 hours) analysis of variance with repeated measures on the third factor. Data presented here are for the drug * time interaction; Test type: Superiority or Other; p = 0.98, ANOVA — P < 0.05 considered statistically significant; Adjustments to the degrees of freedom were made when assumptions of sphericity were violated

2. Secondary Outcome: Change in High Altitude Headache by Visual Analogue Scale
Description: Baseline is defined as the average of the 3 hour and 12 hour normoxia measurement. 24 hours is defined at the 24 hour hypoxia measurement. Outcome measured using visual analogue scale, where 0 mm is no headache and 100 mm is maximum headache.
Time Frame: High Altitude Headache: baseline, 24 hours.
Population: All participants were included. Analysis was intention to treat. There were no missing data.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 11 | 12
mm | 6.4 (10.5) | 7.2 (10.5)
Statistical Analysis 1: Comparison: Acetazolamide vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.63, ANOVA — P < 0.05 considered statistically significant; Adjustments to the degrees of freedom were made when assumptions of sphericity were violated

3. Secondary Outcome: Change in Blood Oxygen Saturation
Description: Baseline is defined as the average of the 3 hour and 12 hour normoxia measurement. 24 hours is defined at the 24 hour hypoxia measurement.
Time Frame: Blood Oxygen Saturation: baseline, 24 hours.
Population: All participants were included. Analysis was intention to treat. There were no missing data.
Measure: Mean (Standard Deviation); unit: % oxygen saturation
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 11 | 12
% oxygen saturation | 10.8 (4.3) | 11.1 (4.3)
Statistical Analysis 1: Comparison: Acetazolamide vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.20, ANOVA — P < 0.05 considered statistically significant; Adjustments to the degrees of freedom were made when assumptions of sphericity were violated

4. Secondary Outcome: Change in Fluid Balance
Description: Baseline is defined as the average of the 3 hour and 12 hour normoxia measurement. 24 hours is defined at the 24 hour hypoxia measurement. Urine output was recorded by 24 hour urine collection and fluid intake by 24 hour food diaries. Fluid balance was calculated as:
  (urine output (L) / fluid intake (L) ) * 100.
Time Frame: Fluid Balance: baseline, 24 hours.
Population: All participants were included. Analysis was intention to treat. There were no missing data.
Measure: Mean (Standard Deviation); unit: % of fluid intake
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 11 | 12
% of fluid intake | 342 (109) | 147 (85)
Statistical Analysis 1: Comparison: Acetazolamide vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.01, ANOVA — P < 0.05 considered statistically significant; Adjustments to the degrees of freedom were made when assumptions of sphericity were violated
Statistical Analysis 2: Comparison: Acetazolamide vs Placebo; Post hoc follow up test. T test between acetazolamide and placebo on data at 24 hr time point; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — Step down Holm Bonferroni correction was applied

5. Secondary Outcome: Change in Optic Nerve Sheath Diameter
Description: Baseline is defined as the average of the 3 hour 12 hour normoxia measurements. 3 hours is defined at the 3 hour hypoxia measurement.
Time Frame: Optic Nerve Sheath Diameter: baseline, 3 hours.
Population: All participants were included. Analysis was intention to treat. There were no missing data.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 11 | 12
mm | 0.00 (0.06) | -0.01 (0.06)
Statistical Analysis 1: Comparison: Acetazolamide vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.98, ANOVA — P < 0.05 considered statistically significant; Adjustments to the degrees of freedom were made when assumptions of sphericity were violated

6. Secondary Outcome: Change in Optic Nerve Sheath Diameter
Description: Baseline is defined as the average of the 3 hour 12 hour normoxia measurements. 12 hours is defined at the 12 hour hypoxia measurement.
Time Frame: Optic Nerve Sheath Diameter: baseline, 12 hours.
Population: All participants were included. Analysis was intention to treat. There were no missing data.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 11 | 12
mm | 0.01 (0.04) | 0.01 (0.04)
Statistical Analysis 1: Comparison: Acetazolamide vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.98, ANOVA — P < 0.05 considered statistically significant; Adjustments to the degrees of freedom were made when assumptions of sphericity were violated

7. Secondary Outcome: Change in Optic Nerve Sheath Diameter
Description: Baseline is defined as the average of the 3 hour and 12 hour normoxia measurements. 36 hours is defined at the 36 hour hypoxia measurement.
Time Frame: Optic Nerve Sheath Diameter: baseline, 36 hours.
Population: All participants were included. Analysis was intention to treat. There were no missing data.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 11 | 12
mm | 0.01 (0.04) | 0.00 (0.04)
Statistical Analysis 1: Comparison: Acetazolamide vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.98, ANOVA — P < 0.05 considered statistically significant; Adjustments to the degrees of freedom were made when assumptions of sphericity were violated

ADVERSE EVENTS:
Time Frame: Study data collection period only (baseline and high altitude exposures up to 36 hours).
Description: Adverse events recorded by study investigators at six hourly interviews.
Arm/Group | Acetazolamide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12

LIMITATIONS AND CAVEATS:
Acetazolamide did not reduce high altitude headache as expected. Nevertheless the relationship between optic nerve sheath diameter and headache could still be determined by completing other analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes